CLINICAL TRIAL: NCT03865589
Title: Using Ultrasound Elastography to Predict Development of Hepatic Sinusoidal Obstruction Syndrome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: Jazz Pharmaceuticals (Industry); Nationwide Children's Hospital (Other); Dana-Farber Cancer Institute (Other); University of California, San Francisco (Other); University Hospitals Cleveland Medical Center (Other); Duke University (Other)
Responsible Party: Principal Investigator, Sherwin Chan MD PhD, Physician, MD, PhD, Children's Mercy Hospital Kansas City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY0000548
Record Dates: First submitted 2019-03-01; First posted 2019-03-07 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Bone Marrow Transplant Complications; Sinusoidal Obstruction Syndrome; Veno Occlusive Disease, Hepatic; Stem Cell Transplant Complications
Keywords: Ultrasound Elastography
MeSH Terms: conditions — Hepatic Veno-Occlusive Disease

STUDY DESIGN:
Intervention Model Description: All patients undergoing myeloblative conditioning regimen as part of hematopoietic cell transplant will be consecutively studied
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Patients Undergoing HCT (Experimental): All patients enrolled will undergo US SWE at specific time points as outlined in the protocol based on disease course.
  Interventions: Diagnostic Test: Ultrasound Elastography

INTERVENTIONS:
Diagnostic Test: Ultrasound Elastography — Ultrasound shear wave elastography

SUMMARY:
To perform an receiver operating characteristic (ROC) analysis, define a threshold and quantify the sensitivity and specificity of US SWE for risk stratification of patients into three categories as defined by the European Bone Marrow Transplant (EBMT) adult and pediatric criteria: no sinusoidal obstruction syndrome (SOS), mild to moderate SOS, and severe to very severe SOS. Secondarily, the investigators would also like to quantify the temporal relationship between US SWE changes and SOS diagnosis according to various clinical criteria (Modified Seattle, Baltimore, EBMT consortium).

DETAILED DESCRIPTION:
Hepatic sinusoidal obstructive syndrome (SOS), also known as veno-occlusive disease, is a complication of hematopoietic stem cell transplant (HCT) that is associated with high morbidity and mortality. 57,000 patients in the United States and Europe undergo HCT annually and SOS affects up to 15% of these patients. SOS pathogenesis is thought to be caused by damage to the hepatic venous endothelium due to the preparative regimen used before HCT. This damage results in obstruction of blood flow through the liver. Pathology shows collagen deposition in the sinusoids and fibrosis of venous lumens. The severity of the disease is not correlated to the number and severity of the histological changes. Mild and moderate SOS can resolve with supportive treatment. Severe SOS (30% of SOS) is commonly associated with multi-organ failure and has a mortality rate of 80% despite available prophylaxis and treatment.

SOS is most commonly defined by two clinical criteria: the modified Seattle criteria and the Baltimore criteria. The modified Seattle criteria state that at least two of the following criteria must be present within 20 days of HCT: bilirubin > 2mg/dL; hepatomegaly and/or ascites; and/or weight gain > 5% above baseline weight (6). Pediatric SOS incidence in HCT is 20% and is higher compared to adults. Death or multi-organ dysfunction affects 30-60% children who develop SOS. The most common definition of severe SOS is retrospective, namely death from SOS-related causes or persistent multi-organ dysfunction at 100 days post HCT. However, the European Society for Blood and Marrow Transplantation has proposed new prospective SOS diagnosis and grading schemes that could become standard of care since it can be performed prospectively and thus can guide treatment.

Defibrotide is a DNA derivative from porcine intestine that protects and repairs endothelial cells. Prior trials showed that defibrotide decreased the incidence of multi-organ failure and death from SOS. The main caveat is that treatment must be initiated very close to the time of clinical diagnosis using the Baltimore criteria to be effective (14). A study showed that 31/33 (94%) patients had complete remission of their SOS when treated with defibrotide <3 days after diagnosis, whereas only 3/12 (25%) patients had complete remission when treated >3 days of diagnosis. However, universal prophylaxis is difficult due to high drug costs ($155,000 for 21-day course). There is a critical need for an early and effective SOS diagnostic test that can identify patients who would benefit from defibrotide treatment.

Several adult and pediatric prospective studies have evaluated the efficacy of grayscale and Doppler ultrasound (US) in diagnosing SOS and have concluded that the clinical criteria are superior to US criteria for SOS diagnosis. The main reason for this conclusion is that conventional US is able to diagnose SOS only after the clinical diagnosis. This research has resulted in multiple recent guidelines recommending US only for confirming clinical diagnoses or following disease progression and not for primary diagnosis. Ultrasound shear wave elastography (SWE) has been shown to effectively diagnose passive hepatic congestion. Fontan physiology is the best studied example. SWE values markedly increased after the Fontan operation. This surgery connects the hepatic venous circulation to the pulmonary arteries exposing the liver to increased resistance from the pulmonary circulation thereby increasing hepatic venous congestion. Additionally, the effect sizes in the Fontan studies are large compared with the effect sizes in hepatic fibrosis studies. The common thread of hepatic venous congestion between Fontan physiology and SOS physiology led us to hypothesize that SWE could be useful in SOS diagnosis. Additionally, preliminary SWE studies in adults showed that it might be useful in the setting of SOS.

The investigators of this study recently conducted a single site prospective cohort study involving 25 patients undergoing myeloablative HCT patients from December 2015 through June 2017. The investigators found increased velocities in all patients who developed SOS. US SWE velocity values showed no difference between pre-conditioning median US SWE velocity in the SOS group (1.24 + 0.09 m/s) and non-SOS group (1.41 + 0.18 m/s) (p=0.06). By day +5, patients with SOS had US SWE velocities that significantly increased by 0.25 + 0.21 m/s from baseline compared to 0.02 + 0.18 m/s in patients without SOS from baseline (p=0.02). By day +14, patients with SOS had US SWE velocities that significantly increased by 0.91 + 1.14 m/s from baseline compared to 0.03 + 0.23 m/s in patients without SOS from baseline (0.01). These values are both clinically and statistically significant, demonstrating that patients with SOS have significantly increased liver stiffness as measured by US SWE compared to patients without SOS. Additionally, SWE changes happened on average 9 to 11 days before clinical diagnostic criteria became positive. The sensitivity and specificity of this test were 60-80% and 67-93% in our small cohort of 25 patients depending on the threshold used and the test timing.

Data Collection Procedures: Candidates for the study will be identified by a HCT physician taking care of the patient and will be identified as a potential candidate for the study. Subjects will be approached for consent by a member of the research team prior to start of conditioning regimen. Consented subjects will have demographic, laboratory and clinical data collected from the chart at each ultrasound time point.

Consented subjects will have an US SWE within two weeks prior to starting their conditioning regimen and at the following time points based on disease course:

1. All Patients: patients will undergo ultrasound elastography within two-weeks prior to admission for conditioning AND twice per week through Day +30 or discharge, whichever comes first.

   Patients whom are still an inpatient after Day +30, and are not clinically suspicious for SOS/VOD, will undergo ultrasound elastography every 30 days (Day +60 and Day +90) until discharge.
2. Late Onset SOS/VOD as INPATIENT (AFTER DAY +30): patients will undergo ultrasound elastography twice a week during course of SOS/VOD treatment. If patient is still admitted at end of treatment, patient will undergo ultrasound elastography once every 30 days through day +100 or discharge, whichever comes first.
3. Late Onset SOS/VOD as OUTPATIENT (DAY +30 - DAY + 100): patients will undergo ultrasound elastography once a week during course of SOS/VOD treatment

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing a myeloablative conditioning regimen for HCT between 3/1/2019 and 12/31/2025 defined as one of the following:

  * TBI >= 1200 cGy (fractionated)
  * Cyclophosphamide + TBI (> 500 cGy (single) or > 800cGy (fractionated))
  * Cyclophosphamide + Etoposide + TBI (> 500 cGy (single) or > 800 cGy (fractionated))
  * Cyclophosphamide + Thiotepa + TBI (> 500 cGy (single) or > 800 cGy (fractionated))
  * Busulfan (Total dose > 7.2 mg/kg IV or >9.0mg/kg orally) + Cyclophosphamide
  * Busulfan (Total dose >7.2 mg/kg IV or >9.0 mg/kg orally) + Melphalan
  * Busulfan (Total dose >7.2 mg/kg IV or >9.0 mg/kg orally) + Thiotepa
  * NOTE: Busulfan cumulative plasma AUC of >75 mg/L per hour or >18270 microMolar per minute could be used in the preceding criteria in lieu of the mg/kg doses.

OR

2. Any patient who has a myeloablative conditioning regimen (as defined by the local HCT team) that includes sirolimus and tacrolimus for GVHD prophylaxis.

OR

3. Any patient who is high risk for SOS irrespective of conditioning regimen: Neuroblastoma, HLH, Osteopetrosis, Thalassemia, treatment with inotuzumab or gemtuzumab within 3 months prior to HCT admission, 2nd HCT if it is myeloablative and within 6 months of prior, iron overload, steatohepatitis, active inflammatory or infection hepatitis or any other condition which puts the patient at a higher risk of developing SOS.

Subjects aged 1 month through 99 years will be eligible for the study. Patients who receive defibrotide and/or ursodiol for VOD/SOS prophylaxis will also be eligible for the study. At most 175 children (ages 1 month to 18 years) and 175 adults (>18 years old) can be enrolled into the study.

Inclusion dates: Patients seen between 1/1/2019 and 12/31/2025

Exclusion Criteria:

Any patient who has contraindication to ultrasound shear wave elastography (e.g. unable to hold still) Adults unable to consent Pregnant women Prisoners Wards of the state

Ages: 1 Month to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Define Sensitivity and Specificity Threshold for US SWE Risk | 100 days post transplant
  To define a threshold and quantify the sensitivity and specificity of US SWE for risk stratification of patients into three categories as defined by the EBMTC adult and pediatric criteria: no SOS, mild to moderate SOS, and severe to very severe SOS

SECONDARY OUTCOMES:
Quantify Temporal Relationship between SWE and SOS and Modified Seattle Criteria | 100 days post transplant
  Quantify the temporal relationship between US SWE changes and SOS diagnosis according to Modified Seattle Criteria
Quantify Temporal Relationship between SWE and SOS and Baltimore Criteria | 100 days post transplant
  Quantify the temporal relationship between US SWE changes and SOS diagnosis according to various clinical criteria Baltimore Criteria
Quantify Temporal Relationship between SWE and SOS and EBMT Consortium | 100 days post transplant
  Quantify the temporal relationship between US SWE changes and SOS diagnosis according to EBMT consortium.

CONTACTS AND LOCATIONS:
Overall Officials: Sherwin S Chan, MD, PhD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (7):
- United States (7):
  - University of California, San Francisco, San Francisco, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Children's Mercy, Kansas City, Missouri
  - Duke University, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - St. Jude Children's Research Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] B. Cozadd, paper presented at the 36th Annual J.P. Morgan Annual Healthcare Conference, San Francisco, California, January 8, 2018 2018
- [Background] Z. X. D'Souza A. (Available at: http://www.cibmtr.org, 2016), vol. 2017
- [Background] P. Negrin RS; Bonis, M. Nelson J Chao, Ed. (www.uptodate.com, 2017), vol. 2017
- [Background] Shulman HM, Fisher LB, Schoch HG, Henne KW, McDonald GB. Veno-occlusive disease of the liver after marrow transplantation: histological correlates of clinical signs and symptoms. Hepatology. 1994 May;19(5):1171-81. PMID 8175139
- [Background] Mohty M, Malard F, Abecassis M, Aerts E, Alaskar AS, Aljurf M, Arat M, Bader P, Baron F, Bazarbachi A, Blaise D, Ciceri F, Corbacioglu S, Dalle JH, Dignan F, Fukuda T, Huynh A, Masszi T, Michallet M, Nagler A, NiChonghaile M, Okamoto S, Pagliuca A, Peters C, Petersen FB, Richardson PG, Ruutu T, Savani BN, Wallhult E, Yakoub-Agha I, Duarte RF, Carreras E. Revised diagnosis and severity criteria for sinusoidal obstruction syndrome/veno-occlusive disease in adult patients: a new classification from the European Society for Blood and Marrow Transplantation. Bone Marrow Transplant. 2016 Jul;51(7):906-12. doi: 10.1038/bmt.2016.130. Epub 2016 May 16. PMID 27183098
- [Background] McDonald GB, Hinds MS, Fisher LD, Schoch HG, Wolford JL, Banaji M, Hardin BJ, Shulman HM, Clift RA. Veno-occlusive disease of the liver and multiorgan failure after bone marrow transplantation: a cohort study of 355 patients. Ann Intern Med. 1993 Feb 15;118(4):255-67. doi: 10.7326/0003-4819-118-4-199302150-00003. PMID 8420443
- [Background] Jones RJ, Lee KS, Beschorner WE, Vogel VG, Grochow LB, Braine HG, Vogelsang GB, Sensenbrenner LL, Santos GW, Saral R. Venoocclusive disease of the liver following bone marrow transplantation. Transplantation. 1987 Dec;44(6):778-83. doi: 10.1097/00007890-198712000-00011. PMID 3321587
- [Background] Corbacioglu S, Cesaro S, Faraci M, Valteau-Couanet D, Gruhn B, Rovelli A, Boelens JJ, Hewitt A, Schrum J, Schulz AS, Muller I, Stein J, Wynn R, Greil J, Sykora KW, Matthes-Martin S, Fuhrer M, O'Meara A, Toporski J, Sedlacek P, Schlegel PG, Ehlert K, Fasth A, Winiarski J, Arvidson J, Mauz-Korholz C, Ozsahin H, Schrauder A, Bader P, Massaro J, D'Agostino R, Hoyle M, Iacobelli M, Debatin KM, Peters C, Dini G. Defibrotide for prophylaxis of hepatic veno-occlusive disease in paediatric haemopoietic stem-cell transplantation: an open-label, phase 3, randomised controlled trial. Lancet. 2012 Apr 7;379(9823):1301-9. doi: 10.1016/S0140-6736(11)61938-7. Epub 2012 Feb 23. PMID 22364685
- [Background] Barker CC, Butzner JD, Anderson RA, Brant R, Sauve RS. Incidence, survival and risk factors for the development of veno-occlusive disease in pediatric hematopoietic stem cell transplant recipients. Bone Marrow Transplant. 2003 Jul;32(1):79-87. doi: 10.1038/sj.bmt.1704069. PMID 12815482
- [Background] Cesaro S, Pillon M, Talenti E, Toffolutti T, Calore E, Tridello G, Strugo L, Destro R, Gazzola MV, Varotto S, Errigo G, Carli M, Zanesco L, Messina C. A prospective survey on incidence, risk factors and therapy of hepatic veno-occlusive disease in children after hematopoietic stem cell transplantation. Haematologica. 2005 Oct;90(10):1396-404. PMID 16219577
- [Background] Coppell JA, Richardson PG, Soiffer R, Martin PL, Kernan NA, Chen A, Guinan E, Vogelsang G, Krishnan A, Giralt S, Revta C, Carreau NA, Iacobelli M, Carreras E, Ruutu T, Barbui T, Antin JH, Niederwieser D. Hepatic veno-occlusive disease following stem cell transplantation: incidence, clinical course, and outcome. Biol Blood Marrow Transplant. 2010 Feb;16(2):157-68. doi: 10.1016/j.bbmt.2009.08.024. Epub 2009 Sep 18. PMID 19766729
- [Background] Richardson PG, Soiffer RJ, Antin JH, Uno H, Jin Z, Kurtzberg J, Martin PL, Steinbach G, Murray KF, Vogelsang GB, Chen AR, Krishnan A, Kernan NA, Avigan DE, Spitzer TR, Shulman HM, Di Salvo DN, Revta C, Warren D, Momtaz P, Bradwin G, Wei LJ, Iacobelli M, McDonald GB, Guinan EC. Defibrotide for the treatment of severe hepatic veno-occlusive disease and multiorgan failure after stem cell transplantation: a multicenter, randomized, dose-finding trial. Biol Blood Marrow Transplant. 2010 Jul;16(7):1005-17. doi: 10.1016/j.bbmt.2010.02.009. Epub 2010 Feb 16. PMID 20167278
- [Background] Corbacioglu S, Carreras E, Ansari M, Balduzzi A, Cesaro S, Dalle JH, Dignan F, Gibson B, Guengoer T, Gruhn B, Lankester A, Locatelli F, Pagliuca A, Peters C, Richardson PG, Schulz AS, Sedlacek P, Stein J, Sykora KW, Toporski J, Trigoso E, Vetteranta K, Wachowiak J, Wallhult E, Wynn R, Yaniv I, Yesilipek A, Mohty M, Bader P. Diagnosis and severity criteria for sinusoidal obstruction syndrome/veno-occlusive disease in pediatric patients: a new classification from the European society for blood and marrow transplantation. Bone Marrow Transplant. 2018 Feb;53(2):138-145. doi: 10.1038/bmt.2017.161. Epub 2017 Jul 31. PMID 28759025
- [Background] Corbacioglu S, Greil J, Peters C, Wulffraat N, Laws HJ, Dilloo D, Straham B, Gross-Wieltsch U, Sykora KW, Ridolfi-Luthy A, Basu O, Gruhn B, Gungor T, Mihatsch W, Schulz AS. Defibrotide in the treatment of children with veno-occlusive disease (VOD): a retrospective multicentre study demonstrates therapeutic efficacy upon early intervention. Bone Marrow Transplant. 2004 Jan;33(2):189-95. doi: 10.1038/sj.bmt.1704329. PMID 14661036
- [Background] The Medical Letter. (https://secure.medicalletter.org/w1503c, 2016), vol. 2017.
- [Background] McCarville MB, Hoffer FA, Howard SC, Goloubeva O, Kauffman WM. Hepatic veno-occlusive disease in children undergoing bone-marrow transplantation: usefulness of sonographic findings. Pediatr Radiol. 2001 Feb;31(2):102-5. doi: 10.1007/s002470000373. PMID 11214676
- [Background] Hommeyer SC, Teefey SA, Jacobson AF, Higano CS, Bianco JA, Colacurcio CJ, McDonald GB. Venocclusive disease of the liver: prospective study of US evaluation. Radiology. 1992 Sep;184(3):683-6. doi: 10.1148/radiology.184.3.1509050.
- [Background] Teefey SA, Brink JA, Borson RA, Middleton WD. Diagnosis of venoocclusive disease of the liver after bone marrow transplantation: value of duplex sonography. AJR Am J Roentgenol. 1995 Jun;164(6):1397-401. doi: 10.2214/ajr.164.6.7754881.
- [Background] Bajwa RPS, Mahadeo KM, Taragin BH, Dvorak CC, McArthur J, Jeyapalan A, Duncan CN, Tamburro R, Gehred A, Lehmann L, Richardson P, Auletta JJ, Woolfrey AE. Consensus Report by Pediatric Acute Lung Injury and Sepsis Investigators and Pediatric Blood and Marrow Transplantation Consortium Joint Working Committees: Supportive Care Guidelines for Management of Veno-Occlusive Disease in Children and Adolescents, Part 1: Focus on Investigations, Prophylaxis, and Specific Treatment. Biol Blood Marrow Transplant. 2017 Nov;23(11):1817-1825. doi: 10.1016/j.bbmt.2017.07.021. Epub 2017 Jul 25. PMID 28754544
- [Background] Kutty SS, Peng Q, Danford DA, Fletcher SE, Perry D, Talmon GA, Scott C, Kugler JD, Duncan KF, Quiros-Tejeira RE, Kutty S; Liver Adult-Pediatric-Congenital-Heart-Disease Dysfunction Study (LADS) Group. Increased hepatic stiffness as consequence of high hepatic afterload in the Fontan circulation: a vascular Doppler and elastography study. Hepatology. 2014 Jan;59(1):251-60. doi: 10.1002/hep.26631. Epub 2013 Nov 19. PMID 23913702
- [Background] Dillman JR, Heider A, Bilhartz JL, Smith EA, Keshavarzi N, Rubin JM, Lopez MJ. Ultrasound shear wave speed measurements correlate with liver fibrosis in children. Pediatr Radiol. 2015 Sep;45(10):1480-8. doi: 10.1007/s00247-015-3345-5. Epub 2015 Apr 8. PMID 25851300
- [Background] Karlas T, Weber J, Nehring C, Kronenberger R, Tenckhoff H, Mossner J, Niederwieser D, Troltzsch M, Lange T, Keim V. Value of liver elastography and abdominal ultrasound for detection of complications of allogeneic hemopoietic SCT. Bone Marrow Transplant. 2014 Jun;49(6):806-11. doi: 10.1038/bmt.2014.61. Epub 2014 Apr 7. PMID 24710567
- [Background] Reddivalla N, Robinson AL, Reid KJ, Radhi MA, Dalal J, Opfer EK, Chan SS. Using liver elastography to diagnose sinusoidal obstruction syndrome in pediatric patients undergoing hematopoetic stem cell transplant. Bone Marrow Transplant. 2020 Mar;55(3):523-530. doi: 10.1038/s41409-017-0064-6. Epub 2018 Jan 15. PMID 29335626